CLINICAL TRIAL: NCT05159700
Title: A Phase I, First-In-Human, Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of PRJ1-3024 in Subjects With Advanced Solid Tumors
Brief Title: A Phase I Study, Evaluating the Safety, Pharmacokinetics and Efficacy of PRJ1-3024 in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhuhai Yufan Biotechnologies Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRJ1-3024 CS101
Record Dates: First submitted 2021-12-07; First posted 2021-12-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor; Advanced Solid Malignancies
Keywords: First in human; Maximum tolerated dose; Recommended Phase 2 dose; Dose Escalation; Hematopoietic progenitor kinase 1; PRJ1-3024
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, open label, 3+3 dose escalation study to determine the safety and preliminary efficacy of PRJ1-3024.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Monotherapy Escalation (Experimental): 3+3 Dose escalation arm with PRJ1-3024 which will begin with 2 subjects treated at the lowest planned dose level PRJ1-3024 is administered orally once daily. The starting dose is 80mg/day.
  Interventions: Drug: PRJ1-3024

INTERVENTIONS:
Drug: PRJ1-3024 — PRJ1-3024 is provided as capsules and is administered orally once a day.

SUMMARY:
This is a Phase I, multicenter, open-label, 3+3 dose escalation study to determine the safety and preliminary efficacy of PRJ1-3024 in subjects with relapsed/refractory solid tumors.

DETAILED DESCRIPTION:
The study will evaluate the safety, tolerability, PK, and pharmacodynamics of PRJ1-3024 and will determine the maximum tolerated dose in subjects with advanced solid tumors.

PRJ1-3024 will be evaluated as an oral therapeutic that tests the anti-tumor activity of PRJ1-3024 in patients with solid tumors and has not yet been tested in humans.

This study will find the safe and tolerable recommended dose in subjects with advanced solid tumors as a open-label, 3+3 dose escalation study.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced (unresectable) or metastatic r/r solid tumors for which no standard therapy is available or for whom standard therapy is considered unsuitable or intolerable.
* Male or non-pregnant, non-lactating female subjects age ≥18 years.
* ECOG Performance Status 0~2.
* Has at least 1 measurable lesion as defined by RECIST 1.1 criteria .
* Life expectancy of >3 months, in the opinion of the Investigator.
* Able to take oral medications and willing to record daily adherence to investigational product.
* Adequate hematologic parameters unless clearly due to the disease under study.
* Adequate renal and hepatic function
* Able to understand and willing to sign a written informed consent form.

Key Exclusion Criteria:

* History of another malignancy
* Known symptomatic brain metastases requiring >10 mg/day of prednisolone.
* Significant cardiovascular disease
* Known active HBV, HCV, AIDS-related illness.
* Has received a live vaccine within 30 days
* History of active autoimmune disorders or ongoing immunosuppressive therapy.
* Receiving concurrent anti-cancer therapy, investigational product, strong inhibitors or inducers of cytochrome P450 3A (CYP3A) .
* Prior treatment with hematopoietic progenitor kinase 1 (HPK1) inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) events during the DLT monitoring period | Day 1 to Day 21
  Safety listings and pharmacokinetic listings will be used for evaluation

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | 24 months
  Characterized by type, seriousness, relationship to study treatment, timing, and severity.
Pharmacokinetic parameter： Accumulation ratio | 24 months
  to estimate the accumulation of PRJ1-3024 from time 0 to the time of last quantifiable concentration after multiple administration
Objective response rate (ORR) | 24 months
  estimated by the proportion of subjects having a complete response (CR) or partial response (PR) with use of RECIST v1.1 criteria.
Duration of response (DOR) | 24 months
  defined as time from the first occurrence of a documented objective response to the time of relapse or death from any cause.
Pharmacokinetic parameter：AUC（0-last） | 24 months
  Area under the concentration-time curve AUC from time 0 to the time of the last quantifiable concentration
Pharmacokinetic parameter：Maximum observed concentration (Cmax) | 24 months
  assessed as time from time 0 to the time of the last quantifiable concentration

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xu, PhD, Study Director — Head of US Clinical Development
Locations (6):
- United States (6):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Christ Hospital, Cincinnati, Ohio
  - NEXT Oncology, Austin, Texas
  - Mays Cancer Center, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No